CLINICAL TRIAL: NCT07333443
Title: Caffeine Ingestion at Acute and Moderate Doses Does Not Improve Sport Climbing Performance: Results From a Randomized Controlled Trial.
Brief Title: Caffeine and Sport Climbing Performance
Acronym: Climbing&CAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Alberto Pérez-López, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CEIP/2024/5/117; CEIP/2024/5/117 (Other: CEIP/2024/5/117)
Record Dates: First submitted 2025-12-15; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Climbing; Caffeine
Keywords: sport climbing; grip strength; pull up strength; caffeine; sport performance

STUDY DESIGN:
Intervention Model Description: A triple-blind, randomized, placebo-controlled design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 0 mg/kg of caffeine
  Interventions: Dietary Supplement: Placebo
- Caffeine (Experimental): 3 mg/kg of caffeine
  Interventions: Dietary Supplement: Acute and moderate dose of caffeine (3 mg/kg body mass)

INTERVENTIONS:
Dietary Supplement: Acute and moderate dose of caffeine (3 mg/kg body mass) — Caffeine supplementation was provide to young male climbers.
  Arms: Caffeine
Dietary Supplement: Placebo — Placebo supplementation was provide to young male climbers.
  Arms: Placebo

SUMMARY:
To determine the effects of ingesting caffeine at a dose of 3 mg/kg body mass on pull-up performance and handgrip-related measures in trained climbers.

DETAILED DESCRIPTION:
Introduction: Caffeine is widely recognized as a performance-enhancing substance across numerous athletic disciplines; however, its role in sport climbing has received comparatively limited scientific attention. Because climbing performance relies heavily on grip force, explosive upper-body strength, and localized muscular endurance, this investigation evaluated the short-term impact of a low caffeine dose on climbing-relevant performance outcomes.

Objective: To determine the effects of ingesting caffeine at a dose of 3 mg/kg body mass on pull-up performance and handgrip-related measures in trained climbers.

Methods: Thirteen trained young male climbers participated in a triple-blind, randomized, crossover study design, completing two experimental conditions (caffeine and placebo). Performance assessments included a pull-up one-repetition maximum (1RM), a pull-up power test conducted at multiple external loads, a pull-up endurance test, and several grip performance evaluations, namely maximal dead-hang duration, maximal dead-hang force, and rate of force development (RFD).

ELIGIBILITY:
Inclusion criteria:

* Healthy individuals
* Age between 18 and 40 years
* At least three months of continuous climbing practice
* Ability to hang for at least 5 seconds from an 18-mm edge
* Ability to perform at least one strict body-weight pull-up

Exclusion criteria:

* Any musculoskeletal or medical condition preventing completion of the experimental protocol
* Participation in less than three training sessions per week or a total training volume <150 min/week
* Use of medications or dietary supplements known to affect caffeine metabolism

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Pull-up 1RM | Through study completion, an average of 4 weeks
Pull-up strength and power test 1 | Through study completion, an average of 4 weeks
  Mean and peak velocity will be recorded at 60%, 80%, 90%, 95% and 100% 1RM.
Pull-up strength and power test 2 | Through study completion, an average of 4 weeks
  Mean and peak power will be recorded at 60%, 80%, 90%, 95% and 100%1RM.
Pull-up muscular endurance test | Through study completion, an average of 4 weeks
  Using body mass and perform one set of many repetitions as possible until task failure. The total number of repetitions, Vmean, Vpeak, Wmean and Wpeak were recorded.
Grip endurance in dead-hang. | Through study completion, an average of 4 weeks
  Maximum hanging time (MHT) test at an 18-mm edge depth with each hand
Maximum grip strength in dead-hang | Through study completion, an average of 4 weeks
  using the Strength Test (ST), which measures the maximal external load a participant can sustain for 5 seconds while hanging from an 18-mm edge
Grip rate of force development (RFD). | Through study completion, an average of 4 weeks
  measuring the maximal one-hand pull (voluntary contraction) at an 18 mm edge with a force sensor

SECONDARY OUTCOMES:
Body composition | Through study completion, an average of 4 weeks
  Using bioelectrical impedance
Dietary habits | Through study completion, an average of 4 weeks
  24 h dietary recall
Physical activity habits | Through study completion, an average of 4 weeks
  International Physical Activity Questionnaire (IPAQ)
Rate of perceived exertion | Through study completion, an average of 4 weeks
  Using RPE scale
Mood states | Through study completion, an average of 4 weeks
  Using the Profile of Mood States (POMS) on a 0-4 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Pérez López, PhD, Principal Investigator — University of Alcala
Locations (1):
- Facultad de Medicina y Ciencias de la Salud. Universidad de Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes